CLINICAL TRIAL: NCT04159896
Title: Phase II Multi-Center Trial of ESK981 in Combination With Nivolumab in Patients With Metastatic Castrate Resistant Prostate Cancer
Brief Title: ESK981 and Nivolumab for the Treatment of Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed to accrual on 3/1/21 due to safety concerns since 2 patients experienced CVA events.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-031; P30CA022453 (NIH)
Record Dates: First submitted 2019-10-21; First posted 2019-11-12 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Prostate Carcinoma Metastatic in the Bone; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 11-(2-methylpropyl)-12,13-dihydro-2-methyl-8-(pyrimidin-2-ylamino)-4H-indazolo(5,4-a)pyrrolo(3,4-c)carbazol-4-one; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ESK981, nivolumab) (Experimental): Patients receive ESK981 PO QD for 5 consecutive days per week, followed by a 2-day break. Patients also receive nivolumab IV on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pan-VEGFR/TIE2 Tyrosine Kinase Inhibitor CEP-11981; Biological: Nivolumab

INTERVENTIONS:
Drug: Pan-VEGFR/TIE2 Tyrosine Kinase Inhibitor CEP-11981 — Given PO
  Other Names: 4H-Indazolo(5,4-a)pyrrolo(3,4-C)carbazol-4-one; 2,5,6,11,12,13-Hexahydro-2-methyl-11-(2-methylpropyl)-8-(2-pyrimidinylamino); 856691-93-5; BOL-303213X; CEP 11981; ESK981
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4; BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies the side effects of ESK981 and nivolumab and to see how well they work for the treatment of castration resistant prostate cancer that has spread to other places in the body (metastatic). ESK981 is an investigational drug that targets several important pathways that are believed to play a role in the spread of cancer. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. This study is being done to see if giving ESK981 and nivolumab together works better in treating metastatic castration resistant prostate cancer compared to usual treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the prostate specific antigen (PSA) >= 50% response rate (PSA50) from baseline using the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria to pan-VEGFR/TIE2 tyrosine kinase inhibitor CEP-11981 (ESK981) plus nivolumab in men with metastatic castration resistant prostate cancer (mCRPC) who have progressed on enzalutamide (an oral androgen-receptor inhibitor) and/or abiraterone acetate (an androgen synthesis inhibitor) and chemotherapy (docetaxel and/or cabazitaxel).

II. To assess the safety and tolerability of ESK981 plus nivolumab.

SECONDARY OBJECTIVES:

I. To determine the time to PSA response (TTPR) in patients with mCRPC. II. To determine the duration of PSA response (PRD) in patients with mCRPC. III. To determine PSA progression rates as defined by the PCWG3 criteria. IV. To determine PSA progression free survival (PPFS) as defined by the PCWG3 criteria.

CORRELATIVE/EXPLORATORY/TERTIARY OBJECTIVE:

I. To assess exploratory biomarkers from blood and tumor biopsies.

OUTLINE:

Patients receive ESK981 orally (PO) once daily (QD) for 5 consecutive days per week, followed by a 2-day break. Patients also receive nivolumab intravenously (IV) on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Group (ECOG) performance status =< 1
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v.)5 from toxicities related to any prior treatments, unless adverse event (AE)(s) are clinically non-significant and/or stable on supportive therapy
* Absolute neutrophil count (ANC) >= 1.5 K/mm^3
* Hemoglobin (Hgb) >= 9 g/dL
* Platelets (Plt) >= 100,000/mm^3
* Serum creatinine =< 1.5 times the upper limit of normal OR creatinine clearance > 30 mL/min by Cockcroft-Gault formula
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN with known hepatic metastases)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (=< 5 x ULN with known hepatic metastases)
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) levels =< 1.5 x ULN (If patient is receiving anticoagulation that is expected to alter these levels, should be in targeted therapeutic range for that agent)
* Patient must have progressive disease while receiving androgen deprivation therapy (ADT) defined by any one of the following as per the PCWG3 criteria for PSA, measurable or non-measurable (bone) disease and must have a castrate serum testosterone level (i.e. =< 50 ng/dL) at screening:

  * PSA: At least two consecutive rises in serum PSA, obtained at a minimum of 1-week intervals, with the final value >= 2.0 ng/mL
  * Measurable disease (by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1): >= 20% increase (with an absolute increase of at least 5 mm) in the sum of diameters of all measurable lesions or the development of one or more new lesions. The short axis of a target lymph node must be more than 15 mm to be assessed for change in size
  * Non-measurable (bone) disease: The appearance of two or more new areas of uptake on bone scan consistent with metastatic disease compared to previous imaging during castration therapy. The increased uptake of pre-existing lesions on bone scan will not be taken to constitute progression, and ambiguous results must be confirmed by other imaging modalities (e.g. X-ray, computed tomography [CT] or magnetic resonance imaging [MRI])
* Metastatic prostate cancer (M1) as documented by appropriate medical imaging (i.e. CT-Scan, positron emission tomography [PET] scan or bone scan)
* Progression on a hormonal agent (abiraterone/enzalutamide) and on a chemotherapy agent (docetaxel and/or cabazitaxel) in the metastatic castration resistant setting as per PCWG3 criteria
* Progression on chemotherapy (e.g. docetaxel, cabazitaxel) in the metastatic castration resistant setting. Progression of disease within 6 months of completing docetaxel in the metastatic castrate-sensitive setting is acceptable
* Have signed an informed consent document indicating that the subject understands the purpose of and procedures required for the study and are willing to participate in the study
* Be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Willingness to use contraception by a method that is deemed effective by the investigator throughout the treatment period and for at least 30 days following the last dose of therapy
* Willingness and ability to comply with study procedures and follow-up examination
* Able to swallow and retain oral medication
* Willingness and ability to undergo mandatory tumor biopsy at baseline and at the cycle 3 visit
* Willingness and ability to undergo mandatory whole blood sample collections at baseline, weeks 2-4 in the first cycle, and then monthly

Exclusion Criteria:

* Systemic therapy (other than a gonadotrophin releasing hormone [GnRH] agonist/antagonist) for CRPC within the past two weeks from cycle 1/day 1 including:

  * CYP-17 inhibitors (e.g. ketoconazole, abiraterone)
  * Antiandrogens (e.g. bicalutamide, nilutamide)
  * Second generation antiandrogens (e.g. enzalutamide, ARN-509, galeterone)
  * Immunotherapy (e.g. sipuleucel-T, ipilimumab)
  * Chemotherapy (e.g. docetaxel, cabazitaxel)
* Prior radiopharmaceutical therapy (e.g. radium-223, strontium-89, samarium-153, etc.) within the past year
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements
* The patient is currently on warfarin or heparin therapy
* The patient has any pre-existing coagulopathy, recent hemoptysis, gross hematuria or gastrointestinal bleeding
* The patient has a history of a clinically significant cardiovascular or cerebrovascular event within 3 months prior to study entry
* The patient has uncontrolled hypertension defined as a blood pressure measurement greater than 150 mm Hg systolic or 90 mm Hg diastolic with medication
* The patient has previously been enrolled in the study or received ESK981
* The patient has known hypersensitivity to gelatin or lactose monohydrate
* The patient has taken a medication known to be a potent inducer of CYP1A2, CYP2C8, or CYP3A4 within 4 weeks prior to the first dose of study drug
* Prior treatment with anti-PD/PD-L1/CTLA4/IDO antibody
* Untreated brain metastases or spinal cord compression
* Major surgical procedure or significant traumatic injury within 6 weeks prior to study registration. (> 6 weeks prior to registration is permitted as long as they have fully recovered from any such procedure)
* History of another primary malignancy except for: malignancy treated with curative intent and no known active disease for >= 5 years, adequately treated non-melanoma skin cancer without evidence of disease, adequately treated carcinoma in situ without evidence of disease
* Angina, myocardial infarction symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, percutaneous angioplasty or Coronary arterial bypass surgery within the past 3 months
* The patient has received any investigational drug within 28 days prior to registration or 5 half-lives of the investigational drug, whichever is sooner

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It is a prostate cancer research
Enrollment: 10 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Heath, M.D., Principal Investigator — Barbara Ann Karmanos Institute
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heath EI, Chen W, Choi JE, Dobson K, Smith M, Maj T, Kryczek I, Zou W, Chinnaiyan AM, Qiao Y. Phase II trial of multi-tyrosine kinase inhibitor ESK981 in combination with PD-1 inhibitor nivolumab in patients with metastatic castration-resistant prostate cancer. Invest New Drugs. 2024 Dec;42(6):675-684. doi: 10.1007/s10637-024-01482-8. Epub 2024 Nov 6. PMID 39503807

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a single arm study with run-in phase. All participants, including the run-in phase, received same dose level, so the safety or efficacy will be analyzed in the total n=10 participants as a single group.
Period: Overall Study
Arm/Group | Treatment (ESK981, Nivolumab)
Started | 10
Completed | 0
Not Completed | 10
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — A transient ischaemic attack | 1

BASELINE CHARACTERISTICS:
Population: This is a single arm study with run-in phase. All participants, including the run-in phase, received same dose level, so the safety or efficacy will be analyzed in the total n=10 participants as a single group.
Arm/Group | Treatment (ESK981, Nivolumab)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 72.5 [61 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline PSA [Median (Full Range); unit: ng/mL] | 153.3 [10 to 1197]

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) >= 50% Response Rate (PSA50)
Description: Will assess PSA decline of >= 50% from baseline (PSA50), using the Prostate Cancer Working Group 3 (PCWG3) criteria. Two-sided Wilson type 95% confidence interval (CI) estimates will be calculated.
Time Frame: From treatment administration up to a maximum duration of 27 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (ESK981, Nivolumab)
Number analyzed (Participants) | 10
percentage of participants | 0 [0 to 0.278]

2. Secondary Outcome: Time to PSA Response (TTPR)
Description: Descriptive statistics of TTPR will be used to summarize the time to PSA response. These descriptives will include N, median, mean, standard deviation (SD), interquartile range (IQR), minimum, and maximum.
Time Frame: From treatment administration up to a maximum duration of 27 months
Population: No PSA response occurred. So, time to PSA response is not applicable.
Arm/Group | Treatment (ESK981, Nivolumab)
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of PSA Response (PRD)
Description: The censored distributions will be summarized with the Kaplan-Meier (K-M) survivorship estimate. A graph of the K-M curve will be generated along with the Hall-Wellner 90% confidence band, and a display of the number of patients at risk at several time points, below the X-axis. Summary statistics (6-month rate, 12-month rate, median, etc.) will be calculated from the K-M life table, each one with its respective 80% CI.
Time Frame: From treatment administration up to a maximum duration of 27 months
Population: No PSA response occurred. So, duration of PSA response is not applicable.
Arm/Group | Treatment (ESK981, Nivolumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Time from start of treatment to death due to any cause.
Time Frame: From treatment administration up to a maximum duration of 27 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Treatment (ESK981, Nivolumab)
Number analyzed (Participants) | 10
month | 9.6 [1.8 to 22.4]

5. Other Pre Specified Outcome: Somatic and Germline Mutations
Description: Will assess the proportion of patients with TP53 mutations, AR amplifications, and ETS-fusions, mutations in the PTENPI3K-AKT pathway as well as germline and somatic events in the DNA repair pathway with exceptional response/resistance to pan-VEGFR/TIE2 tyrosine kinase inhibitor CEP-11981 (ESK981).
Time Frame: From treatment administration up to a maximum duration of 27 months
Population: The study was terminated early. All other pre-specified endpoints were not collected.
Arm/Group | Treatment (ESK981, Nivolumab)
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: ETS/Kinase Gene Fusions
Description: Will assess the proportion of patients with ETS/kinase gene fusions with exceptional response/resistance to ESK981.
Time Frame: From treatment administration up to a maximum duration of 27 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Androgen Receptor (AR) Signaling
Description: Will assess the correlation of AR signaling as a predictor of exceptional response to ESK981.
Time Frame: From treatment administration up to a maximum duration of 27 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Metastatic Kinome Activity Profiles as Predictive Biomarkers for Response to ESK981
Description: Will assess the correlation of Metastatic kinome activity profiles as a predictor for exceptional response to ESK981
Time Frame: From treatment administration up to a maximum duration of 27 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Circulating and Disseminated Tumor Cells as Pharmacodynamic Biomarkers of ESK981 Response
Description: Will assess the correlation of circulating and disseminated tumor cells as a predictor for exceptional response to ESK981 .
Time Frame: From treatment administration up to a maximum duration of 27 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Pathological Assessment of Phenotypic Tumor and Host Responses to ESK981 Treatment
Description: Will assess the correlation of IHC % staining as a predictor for exceptional response to ESK981 .
Time Frame: From treatment administration up to a maximum duration of 27 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From treatment administration to 30 days after off-treatment date, up to a maximum of 27 months. Every participant could have different AE observation duration. Patient receives treatment until one of the following off-treatment event occurs: disease progression, toxicity, investigator decision, or patient withdraw.
Description: An adverse event for the purposes of this protocol is the appearance of (or worsening of any pre-existing) undesirable sign, symptom, or medical condition occurring after signing the informed consent even if the event is not considered to be related to the study drug. Every participants in this study, including the safety run-in phase cohort, received same dose level. The AEs will be reported in one group.
Arm/Group | Treatment (ESK981, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 9/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (ESK981, Nivolumab) (N=10)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (ESK981, Nivolumab) (N=10)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (7)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Pain (General disorders) | 6 (10)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Creatinine increased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT04159896/Prot_SAP_000.pdf